CLINICAL TRIAL: NCT00782769
Title: A Multicenter, Parallel-Group Extension Study to Evaluate the Safety of Two Doses of DR-3001 in Women With Overactive Bladder
Brief Title: A Safety Extension Study of DR-OXY-301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-OXY-302
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxybutinyn Vaginal Ring 4mg (Experimental): inserted daily and replaced every 4 weeks
  Interventions: Drug: Oxybutinyn Vaginal Ring 4mg
- Oxybutinyn Vaginal Ring 6mg (Experimental): inserted daily and replaced every 4 weeks
  Interventions: Drug: Oxybutinyn Vaginal Ring 6mg

INTERVENTIONS:
Drug: Oxybutinyn Vaginal Ring 4mg
  Other Names: DR-3001
  Arms: Oxybutinyn Vaginal Ring 4mg
Drug: Oxybutinyn Vaginal Ring 6mg
  Other Names: DR-3001
  Arms: Oxybutinyn Vaginal Ring 6mg

SUMMARY:
This is a safety extension study of DR-OXY-301 at pre-selected sites. Subjects who complete the DR-OXY-301 study are eligible to participate. The duration of this extension study will be up to approximately 42 weeks. Subjects will have physical and laboratory exams, including blood draws at each scheduled visit and colposcopic examination of the vagina and cervix. As in DR-OXY-301, subjects will be required to insert a vaginal ring; replacing it every 4 weeks. Subjects will also be required to keep a daily record of the number of times and the total amount of time the ring was outside the body each day and the reason for voluntary removal.

ELIGIBILITY:
Inclusion Criteria:

* Completed the 12 weeks of treatment in the DR-OXY-301 study
* Willing to limit medications for overactive bladder to investigational product only
* Able to understand and complete all study procedures including the required diary

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety, by investigating post void residual volume, physical exams, vital signs, and clinical laboratory values. The outcome of any pregnancy will be followed and reported | Duration of Study

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Research Protocol Chair, Study Chair — Duramed Research, Inc
Locations (31):
- United States (31):
  - Duramed Investigational Site, Phoenix, Arizona
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, Miami, Florida
  - Duramed Investigational Site, Tampa, Florida
  - Duramed Investigational Site, Augusta, Georgia
  - Duramed Investigational Site, Savannah, Georgia
  - Duramed Investigational Site, Boise, Idaho
  - Duramed Investigational Site, Chicago, Illinois
  - Duramed Investigational Site, Wichita, Kansas
  - Duramed Investigational Site, Louisville, Kentucky
  - Duramed Investigational Site, Watertown, Massachusetts
  - Duramed Investigational Site, Las Vegas, Nevada
  - Duramed Investigational Site, Moorestown, New Jersey
  - Duramed Investigational Site, Albuquerque, New Mexico
  - Duramed Investigational Site, Port Jefferson, New York
  - Duramed Investigational Site, New Bern, North Carolina
  - Duramed Investigational Site, Oklahoma City, Oklahoma
  - Duramed Investigational Site, Eugene, Oregon
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Pottstown, Pennsylvania
  - Duramed Investigational Site, Columbia, South Carolina
  - Duramed Investigational Site, Hilton Head Island, South Carolina
  - Duramed Investigational Site, Jackson, Tennessee
  - Duramed Investigational Site, Houston, Texas
  - Duramed Investigational Site, Waco, Texas
  - Duramed Investigational Site, Williston, Vermont
  - Duramed Investigational Site, Norfolk, Virginia
  - Duramed Investigational Site, Seattle, Washington
  - Duramed Investigational Site, Tacoma, Washington